CLINICAL TRIAL: NCT03305315
Title: Study of Movement of the Pathological Temporomandibular Joint.
Brief Title: Study of Temporomandibular Joint Dysfunction
Acronym: CinématiqueATM
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Other Study IDs: ZWETYENGA ENIM 2016
Record Dates: First submitted 2017-10-04; First posted 2017-10-09 (Actual); Last update posted 2021-01-26 (Actual); Status verified 2021-01

CONDITIONS: Diseases of the Temporomandibular Joint

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cases: Diseases of the temporomandibular joint
  Interventions: Other: Measurements of jaw movement; Other: Measurement of natural electrical activity of facial muscles
- Controls: Asymptomatic subjects
  Interventions: Other: Measurement of natural electrical activity of facial muscles

INTERVENTIONS:
Other: Measurements of jaw movement — Jaw mobility will be measured during simple movements of the mouth (opening the mouth, side-to-side and backwards-and-forwards movement of the jaw). These movements will be measured using a specific apparatus, part of which will be placed on the head like a helmet with the other part placed in the mouth and stuck to the teeth using a dental adhesive. The part in the mouth is specifically designed for this purpose. Measurements using this apparatus will take around 30 minutes.
  Groups: Cases
Other: Measurement of natural electrical activity of facial muscles — Natural electrical activity of the facial muscles will be measured using electrodes placed on the skin.

SUMMARY:
Given the frequency of temporomandibular joint (TMJ) dysfunction and the variations in its expression, this project intends to initiate a process of objective evaluation of mandible function and its impairment due to different diseases. The first step is to determine whether 3D kinematic quantification of the mandible would make it possible to objectively assess the effect of post-operative management on TMJ function recovery. If the first results are encouraging and show the sensitivity of the analysis of minor joint dysfunctions, the investigators will evaluate the feasibility of kinematic assessments for major TMJ dysfunctions and for the follow-up of patients.

The expected benefits of this study are to be considered in the medium term and concern the possibilities offered by measuring mandible kinetics in the treatment of TMJ disorders.

ELIGIBILITY:
Inclusion Criteria:

Patients:

* Patients who have provided verbal consent,
* Patients over 18 years old,
* Patients with mandible dentition compatible with placement of the kinetic measurement device,
* Patients with a TMJ disease requiring surgery (irreducible dislocation of the joint disc, damage to the joint disc requiring discectomy, ankylosis or severe arthritis of the mandible requiring mandible implants or a TMJ prosthesis).

Asymptomatic subjects:

* Subjects who have provided verbal consent,
* Subjects over 18 years old,
* Subjects with Class 1 occlusion,
* Subjects without dental implants,
* Subjects with no history of joint dysfunction,
* Absence of clicking, popping, or grating sounds during large movements and during palpation of the TMJ with the mouth slightly open (distance between incisors around 1 cm)
* Absence of headache,
* Absence of tinnitus,
* Kinematic curves around the mean.

Exclusion Criteria:

* Adults under guardianship,
* Patients without national health insurance cover.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with temporomandibular joint disorders and asymptomatic subjects
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2017-12-12 (Actual); Primary Completion 2019-11-22 (Actual); Study Completion 2019-11-22 (Actual)

PRIMARY OUTCOMES:
Mobility of the jaw with regard to the skull during each movement. | Until 6 months post-surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Dijon Bourogne, Dijon, France